CLINICAL TRIAL: NCT04400929
Title: Using GM-CSF as a Host Directed Therapeutic Against COVID-19 - a Phase 2 Investigator Initiated Trial
Brief Title: Using GM-CSF as a Host Directed Therapeutic Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-Leuk-01
Record Dates: First submitted 2020-05-08; First posted 2020-05-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: COVID; Sars-CoV2; ARDS, Human
Keywords: pandemic; host-directed therapeutic; GM-CSF; COVID-19; ARDS; SARS-CoV2
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled clinical trial of iv Leukine® in 30 patients with confirmed COVID-19 and acute hypoxic respiratory failure.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study to investigate immediate versus delayed treatment of iv Leukine® in improving oxygenation and short- and long-term outcome of COVID-19 patients with acute hypoxic respiratory failure. The study will be unblinded at Day 5, or at any time within the first 5 days of study should the patient deteriorate clinically with need for supplemental oxygen FiO2 requirement ≥ 0.5.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group A: Treatment Group (Experimental): Day 1 - 5: Receive study medication Leukine® 125mcg/m2 body surface area daily (via infusion into the vein) in addition to standard of care treatments
  Interventions: Drug: Sargramostim
- Group B: Placebo Group (Placebo Comparator): Day 1 - 5: Receive normal saline 0.9% daily (via infusion into the vein) in addition to standard of care treatments
  Interventions: Other: Normal Saline 0.9%
- Group C (Experimental): Day 6 - 10: Subjects in Group A who require mechanical ventilation to receive an additional 5 days of IV Leukine® 125mcg/m2 body surface area daily, in addition to standard of care treatments (based on the treating physician's assessment)
  Interventions: Drug: Sargramostim
- Group D (Experimental): Day 6 - 10: Subjects from Group B to receive study medication (based on the treating physician's assessment), Leukine® 125mcg/m2 body surface area daily (via infusion into the vein) in addition to standard of care treatments
  Interventions: Drug: Sargramostim
- Group E (Experimental): Day 11 - 15: Subjects in Group D who require mechanical ventilation to receive an additional 5 days of IV Leukine® 125mcg/m2 body surface area daily, in addition to standard of care treatments (based on the treating physician's assessment)
  Interventions: Drug: Sargramostim

INTERVENTIONS:
Drug: Sargramostim — Dosage for IV Leukine® injection: 125mcg/m2/day over a 4-hour period for up to 5 days.
  Other Names: GM-CSF; Granulocyte-Macrophage Colony Stimulating Factor; Leukine®
  Arms: Group A: Treatment Group; Group C; Group D; Group E
Other: Normal Saline 0.9% — IV normal saline 0.9% for 5 days
  Arms: Group B: Placebo Group

SUMMARY:
The coronavirus disease 2019 (COVID-19) has rapidly become a pandemic. COVID-19 poses a mortality risk of 3-7%, rising to 20% in older patients with co-morbidities. Of all infected patients, 15-20% will develop severe respiratory symptoms necessitating hospital admission. Around 5% of patients will require invasive mechanical ventilation, and up to 50% will die.

Evidence in severe COVID-19 suggests that these patients experience cytokine storm and progressed rapidly with acute respiratory distress syndrome and eventual multi-organ failure. Early identification and immediate treatment of hyperinflammation is thus recommended to reduce mortality. Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) has been shown to be a myelopoietic growth factor that has pleiotropic effects in promoting the differentiation of immature precursors into polymorphonuclear neutrophils, monocytes/ macrophages and dendritic cells, and also in controlling the function of fully mature myeloid cells. It plays an important role in priming monocytes for production of proinflammatory cytokines under TLR and NLR stimulation. It has a broad impact on the processes driving DC differentiation and affects DC effector function at the mature state. Importantly, GM-CSF plays a critical role in host defense and stimulating antiviral immunity. Detailed studies have also shown that GM-CSF is necessary for the maturation of alveolar macrophages from foetal monocytes and the maintenance of these cells in adulthood. The known toxicology, pharmacologic and safety data also support the use of Leukine® in hypoxic respiratory failure and ARDS due to COVID-19.

This study aims to recruit patients with evidence of pneumonia and hypoxia who have increased risk for severe disease and need for mechanical ventilation. The overall hypothesis is that GM-CSF has antiviral immunity, can provide the stimulus to restore immune homeostasis in the lung with acute lung injury from COVID-19, and can promote lung repair mechanisms, which would lead to improvement in lung oxygenation parameters.

DETAILED DESCRIPTION:
The hypothesis of the proposed intervention is that GM-CSF has profound effects on antiviral immunity, can provide the stimulus to restore immune homeostasis in the lung with acute lung injury post COVID-19, and can promote lung repair mechanisms, which would lead to an improvement in lung oxygenation parameters. This hypothesis is based on experiments performed in mice showing that GM-CSF treatment can prevent mortality and prevent ARDS in mice with post-viral acute lung injury.

In the interim analysis of the SARPAC trial, patients who received nebulised Leukine® via a mesh inhaler showed a trend in improvement in their P(A-a)O2 gradient at day 6 compared to the SOC group. There are however, anticipated logistical difficulties of training and infection control concerns with administering of nebulised Leukine® via a specialised inhaler in the negative pressure room. Hence we propose to randomize patients with confirmed COVID-19 and acute hypoxic respiratory failure (saturation < 94% on room air or PaO2/FiO2 <350) to receive iv Leukine® 125mcg/m2 once a day for 5 days on top of SOC (treatment group A), or to receive SOC treatment only (placebo group B). Dosing of systemic Leukine® is based on prior experience of using this drug in patients with pneumonia-associated ARDS.

To measure the effectiveness of Leukine® in restoring lung homeostasis, the primary endpoint of this intervention is measuring oxygenation after 5 days of intravenous treatment through assessment of pre-treatment and post-treatment ratio of PaO2/FiO2, and through measurement of the P(A-a)O2 gradient, which can easily be performed in the setting of clinical observation of inpatients. During the 5-day treatment period, we will perform daily measurements of oxygen saturation (pulse oximetry) in relation to FiO2, and the slope of alterations in these parameters could also be an indicator that our hypothesis is correct.

Comparison will be between group A receiving iv Leukine® on top of standard of care (SOC) and placebo group B receiving SOC only. Data from the Wuhan COVID-19 epidemic show that patients that deteriorate are facing a prolonged period of mechanical ventilation. Therefore, the study will be unblinded at day 5, or at any time within the first 5 days of study should the patient deteriorate clinically with need for supplemental oxygen FiO2 requirement ≥ 0.5. Patients in group B will then have the option to receive 5 days of iv Leukine®, based on the treating physician's assessment. This group will be group D. Patients who require mechanical ventilation also have the option to receive an additional 5 days of iv Leukine®, based on the treating physician's assessment (group C and E).

A total of 30 patients with confirmed COVID-19 and acute hypoxic respiratory failure will be enrolled, 15 who will receive Leukine® + SOC, and 15 who will receive placebo + SOC. The target group of subjects is defined as confirmed COVID-19 patients with acute hypoxic respiratory failure admitted to the COVID-19 isolation ward. Subjects will be recruited from the isolation wards located in Singapore General Hospital (SGH). Subjects will be identified by the primary managing physicians who are infectious diseases physicians.

Safety data, including blood leukocyte counts, will be collected in all patients. Efficacy data will also be collected and will include arterial blood gases, oxygenation parameters, need for ventilation, lung compliance, organ function, radiographic changes, ferritin levels, triglyceride levels, etc. as well as occurrence of secondary bacterial infections.

Patients will stop the investigational drug if there is unacceptable toxicity according to investigator's judgement.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 PCR-confirmed COVID-19 infection
* Presence of acute hypoxic respiratory failure defined as (either or both)
* Saturation < 94% on room air or requiring supplemental oxygen
* PaO2/FiO2 below 350
* Age 21-80
* Able and willing to provide informed consent

Exclusion Criteria:

* Patients who are already on supplemental oxygen of FiO2 ≥ 0.4
* Patients with known history of serious allergic reactions, including anaphylaxis, to human GM-CSF such as Leukine®, yeast-derived products, or any component of the product.
* Mechanical ventilation before start of study
* Patients enrolled in another investigational drug study
* Pregnant or breastfeeding females (all female subjects of childbearing potential status must have negative pregnancy test at screening)
* Patients with peripheral white blood cell count above 25,000 per microliter and/or active myeloid malignancy
* Patients on high dose systemic steroids (> 20mg methylprednisolone or equivalent)
* Patients on lithium carbonate therapy
* Patients with serum ferritin >2000 mcg/ml (which will exclude ongoing HLH)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Measuring oxygenation | Day 1 to Day 6
  To measure the effectiveness of Leukine® in restoring lung homeostasis, the primary endpoint of this intervention is measuring oxygenation after 5 days of intravenous treatment through assessment of pre-treatment and post-treatment ratio of PaO2/FiO2, and through measurement of the P(A-a)O2 gradient, which can easily be performed in the setting of clinical observation of inpatients.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Cheung CY, Poon LL, Ng IH, Luk W, Sia SF, Wu MH, Chan KH, Yuen KY, Gordon S, Guan Y, Peiris JS. Cytokine responses in severe acute respiratory syndrome coronavirus-infected macrophages in vitro: possible relevance to pathogenesis. J Virol. 2005 Jun;79(12):7819-26. doi: 10.1128/JVI.79.12.7819-7826.2005. PMID 15919935
- [Background] Kikkert M. Innate Immune Evasion by Human Respiratory RNA Viruses. J Innate Immun. 2020;12(1):4-20. doi: 10.1159/000503030. Epub 2019 Oct 14. PMID 31610541
- [Background] Prompetchara E, Ketloy C, Palaga T. Immune responses in COVID-19 and potential vaccines: Lessons learned from SARS and MERS epidemic. Asian Pac J Allergy Immunol. 2020 Mar;38(1):1-9. doi: 10.12932/AP-200220-0772. PMID 32105090
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Correction to: Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 Jun;46(6):1294-1297. doi: 10.1007/s00134-020-06028-z. PMID 32253449
- [Background] Park WY, Goodman RB, Steinberg KP, Ruzinski JT, Radella F 2nd, Park DR, Pugin J, Skerrett SJ, Hudson LD, Martin TR. Cytokine balance in the lungs of patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1896-903. doi: 10.1164/ajrccm.164.10.2104013. PMID 11734443
- [Background] Fowler AA, Fisher BJ, Centor RM, Carchman RA. Development of the adult respiratory distress syndrome: progressive alteration of neutrophil chemotactic and secretory processes. Am J Pathol. 1984 Sep;116(3):427-35. PMID 6476079
- [Background] Munford RS, Pugin J. Normal responses to injury prevent systemic inflammation and can be immunosuppressive. Am J Respir Crit Care Med. 2001 Feb;163(2):316-21. doi: 10.1164/ajrccm.163.2.2007102. No abstract available. PMID 11179099
- [Background] Monneret G, Lepape A, Voirin N, Bohe J, Venet F, Debard AL, Thizy H, Bienvenu J, Gueyffier F, Vanhems P. Persisting low monocyte human leukocyte antigen-DR expression predicts mortality in septic shock. Intensive Care Med. 2006 Aug;32(8):1175-83. doi: 10.1007/s00134-006-0204-8. Epub 2006 Jun 2. PMID 16741700
- [Background] Tiegs G, Barsig J, Matiba B, Uhlig S, Wendel A. Potentiation by granulocyte macrophage colony-stimulating factor of lipopolysaccharide toxicity in mice. J Clin Invest. 1994 Jun;93(6):2616-22. doi: 10.1172/JCI117274. PMID 8201000
- [Background] Meisel C, Schefold JC, Pschowski R, Baumann T, Hetzger K, Gregor J, Weber-Carstens S, Hasper D, Keh D, Zuckermann H, Reinke P, Volk HD. Granulocyte-macrophage colony-stimulating factor to reverse sepsis-associated immunosuppression: a double-blind, randomized, placebo-controlled multicenter trial. Am J Respir Crit Care Med. 2009 Oct 1;180(7):640-8. doi: 10.1164/rccm.200903-0363OC. Epub 2009 Jul 9. PMID 19590022
- [Background] Toda H, Murata A, Oka Y, Uda K, Tanaka N, Ohashi I, Mori T, Matsuura N. Effect of granulocyte-macrophage colony-stimulating factor on sepsis-induced organ injury in rats. Blood. 1994 May 15;83(10):2893-8. PMID 8180384
- [Background] Guilliams M, De Kleer I, Henri S, Post S, Vanhoutte L, De Prijck S, Deswarte K, Malissen B, Hammad H, Lambrecht BN. Alveolar macrophages develop from fetal monocytes that differentiate into long-lived cells in the first week of life via GM-CSF. J Exp Med. 2013 Sep 23;210(10):1977-92. doi: 10.1084/jem.20131199. Epub 2013 Sep 16. PMID 24043763
- [Background] Naessens T, Schepens B, Smet M, Pollard C, Van Hoecke L, De Beuckelaer A, Willart M, Lambrecht B, De Koker S, Saelens X, Grooten J. GM-CSF treatment prevents respiratory syncytial virus-induced pulmonary exacerbation responses in postallergic mice by stimulating alveolar macrophage maturation. J Allergy Clin Immunol. 2016 Mar;137(3):700-9.e9. doi: 10.1016/j.jaci.2015.09.031. Epub 2015 Nov 10. PMID 26560044
- [Background] van de Laar L, Saelens W, De Prijck S, Martens L, Scott CL, Van Isterdael G, Hoffmann E, Beyaert R, Saeys Y, Lambrecht BN, Guilliams M. Yolk Sac Macrophages, Fetal Liver, and Adult Monocytes Can Colonize an Empty Niche and Develop into Functional Tissue-Resident Macrophages. Immunity. 2016 Apr 19;44(4):755-68. doi: 10.1016/j.immuni.2016.02.017. Epub 2016 Mar 15. PMID 26992565
- [Background] Presneill JJ, Harris T, Stewart AG, Cade JF, Wilson JW. A randomized phase II trial of granulocyte-macrophage colony-stimulating factor therapy in severe sepsis with respiratory dysfunction. Am J Respir Crit Care Med. 2002 Jul 15;166(2):138-43. doi: 10.1164/rccm.2009005. PMID 12119223
- [Background] Paine R 3rd, Standiford TJ, Dechert RE, Moss M, Martin GS, Rosenberg AL, Thannickal VJ, Burnham EL, Brown MB, Hyzy RC. A randomized trial of recombinant human granulocyte-macrophage colony stimulating factor for patients with acute lung injury. Crit Care Med. 2012 Jan;40(1):90-7. doi: 10.1097/CCM.0b013e31822d7bf0. PMID 21926600
- [Background] Herold S, Hoegner K, Vadasz I, Gessler T, Wilhelm J, Mayer K, Morty RE, Walmrath HD, Seeger W, Lohmeyer J. Inhaled granulocyte/macrophage colony-stimulating factor as treatment of pneumonia-associated acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Mar 1;189(5):609-11. doi: 10.1164/rccm.201311-2041LE. No abstract available. PMID 24579839
- [Background] Tazawa R, Trapnell BC, Inoue Y, Arai T, Takada T, Nasuhara Y, Hizawa N, Kasahara Y, Tatsumi K, Hojo M, Ishii H, Yokoba M, Tanaka N, Yamaguchi E, Eda R, Tsuchihashi Y, Morimoto K, Akira M, Terada M, Otsuka J, Ebina M, Kaneko C, Nukiwa T, Krischer JP, Akazawa K, Nakata K. Inhaled granulocyte/macrophage-colony stimulating factor as therapy for pulmonary alveolar proteinosis. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1345-54. doi: 10.1164/rccm.200906-0978OC. Epub 2010 Feb 18. PMID 20167854
- [Background] Tazawa R, Ueda T, Abe M, Tatsumi K, Eda R, Kondoh S, Morimoto K, Tanaka T, Yamaguchi E, Takahashi A, Oda M, Ishii H, Izumi S, Sugiyama H, Nakagawa A, Tomii K, Suzuki M, Konno S, Ohkouchi S, Tode N, Handa T, Hirai T, Inoue Y, Arai T, Asakawa K, Sakagami T, Hashimoto A, Tanaka T, Takada T, Mikami A, Kitamura N, Nakata K. Inhaled GM-CSF for Pulmonary Alveolar Proteinosis. N Engl J Med. 2019 Sep 5;381(10):923-932. doi: 10.1056/NEJMoa1816216. PMID 31483963
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Halstead ES, Umstead TM, Davies ML, Kawasawa YI, Silveyra P, Howyrlak J, Yang L, Guo W, Hu S, Hewage EK, Chroneos ZC. GM-CSF overexpression after influenza a virus infection prevents mortality and moderates M1-like airway monocyte/macrophage polarization. Respir Res. 2018 Jan 5;19(1):3. doi: 10.1186/s12931-017-0708-5. PMID 29304863
- [Background] Umstead TM, Hewage EK, Mathewson M, Beaudoin S, Chroneos ZC, Wang M, Halstead ES. Lower respiratory tract delivery, airway clearance, and preclinical efficacy of inhaled GM-CSF in a postinfluenza pneumococcal pneumonia model. Am J Physiol Lung Cell Mol Physiol. 2020 Apr 1;318(4):L571-L579. doi: 10.1152/ajplung.00296.2019. Epub 2020 Jan 29. PMID 31994895
- [Background] Rosler B, Herold S. Lung epithelial GM-CSF improves host defense function and epithelial repair in influenza virus pneumonia-a new therapeutic strategy? Mol Cell Pediatr. 2016 Dec;3(1):29. doi: 10.1186/s40348-016-0055-5. Epub 2016 Aug 1. PMID 27480877
- [Background] Zhan Y, Lew AM, Chopin M. The Pleiotropic Effects of the GM-CSF Rheostat on Myeloid Cell Differentiation and Function: More Than a Numbers Game. Front Immunol. 2019 Nov 15;10:2679. doi: 10.3389/fimmu.2019.02679. eCollection 2019. PMID 31803190
- [Background] Schneider C, Nobs SP, Heer AK, Hirsch E, Penninger J, Siggs OM, Kopf M. Frontline Science: Coincidental null mutation of Csf2ralpha in a colony of PI3Kgamma-/- mice causes alveolar macrophage deficiency and fatal respiratory viral infection. J Leukoc Biol. 2017 Feb;101(2):367-376. doi: 10.1189/jlb.4HI0316-157R. Epub 2016 Jul 28. PMID 27468760
- [Background] Unkel B, Hoegner K, Clausen BE, Lewe-Schlosser P, Bodner J, Gattenloehner S, Janssen H, Seeger W, Lohmeyer J, Herold S. Alveolar epithelial cells orchestrate DC function in murine viral pneumonia. J Clin Invest. 2012 Oct;122(10):3652-64. doi: 10.1172/JCI62139. Epub 2012 Sep 10. PMID 22996662
- [Background] Huang FF, Barnes PF, Feng Y, Donis R, Chroneos ZC, Idell S, Allen T, Perez DR, Whitsett JA, Dunussi-Joannopoulos K, Shams H. GM-CSF in the lung protects against lethal influenza infection. Am J Respir Crit Care Med. 2011 Jul 15;184(2):259-68. doi: 10.1164/rccm.201012-2036OC. Epub 2011 Apr 7. PMID 21474645
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533